CLINICAL TRIAL: NCT05481489
Title: Phase I Clinical Trial to Evaluate the Safety and Tolerability of the Ophthalmic Solution PRO-230 When Applied to the Ocular Surface of Healthy Volunteers.
Brief Title: Safety and Tolerability Evaluation of PRO-230 Ophthalmic Solution
Acronym: PRO-230
Status: Withdrawn | Phase: Phase 1 | Type: Interventional
Why Stopped: Due to sponsors convenience.
Sponsor: Laboratorios Sophia S.A de C.V. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: SOPH230-1121/I
Record Dates: First submitted 2022-07-28; First posted 2022-08-01 (Actual); Last update posted 2024-07-01 (Actual); Status verified 2024-06

CONDITIONS: Myopia
MeSH Terms: conditions — Myopia | interventions — Atropine

STUDY DESIGN:
Intervention Model Description: Phase I, non comparative, open, unicentric.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- PRO-230 (Experimental): Healthy volunteers will apply one drop of PRO-230 ophthalmic solution (atropine sulphate) on both eyes, QD (one time per day) for 14 days.
  Interventions: Drug: Atropine Sulfate

INTERVENTIONS:
Drug: Atropine Sulfate — Atropine Sulfate 0.05% Ophthalmic Solution

SUMMARY:
Phase I Study to evaluate safety and tolerability of PRO-230 (atropine sulphate 0.05%) ophthalmic solution through evaluation of incidence of non-expected adverse events (AE), photophobia, pupillary diameter, incidence of expected adverse events, and best near corrected visual acuity (BNCVA)

DETAILED DESCRIPTION:
A total of 29 healthy volunteers will apply PRO-230 ocular solution on both eyes QD (one time per day) for 14 days. The safety variables will include non expected AE, pupillary diameter and expected AE; tolerability variables will include incidence of photofobia, and BNCVA. Exploratory variables include best corrected visual acuity (BCVA), intraocular pressure (IOP), corneal an conjunctival staining with fluorescein and lissamine green, vital signs (heart rate and blood pressure), and results of the Ocular Confort Index (OCI) questionnaire.

The presence of non-expected AE < 10% will deem PRO-230 as safe; while an incidence of photophobia < 30% will deem PRO-230 as tolerable.

ELIGIBILITY:
Inclusion Criteria:

* Being clinically healthy
* Ability to voluntarily sign an informed consent form (ICF).
* Ability and willingness to comply with the scheduled visits according to the intervention plan and other procedures of the study.
* Age between 18 and 35.
* Absence of history of contact lens use.
* Women of childbearing age must agree to continue (starting ≥ 30 days previous to the ICF) the use of a hormonal contraception method of a intrauterine device (IUD) during the period of the study.
* Best corrected visual acuity (BVCA) of at least 20/30 (logMAR 0.2) or better in both eyes.
* Best near corrected visual acuity (BNVCA) of at least 20/25 (logMAR 0.1) or better in both eyes.
* Presenting vital signs within normal parameters.
* Presenting an IOP ≥10 and ≤ 21 mmHg

Exclusion Criteria:

* Using any kind of ophthalmic topical products.
* Presenting known allergy or intolerance to any ingrediente of atropine eyedrops or any other derivatives of antimuscarinic agents.
* Using any medication of herbolary products (plant extracts, infusions, naturist preparations, homeopathy, etc) through any route of administration
* For women: being pregnant, breastfeeding or planning to get pregnant during the period of the study.
* Having participated in any clinical study 90 days prior to the inclusion in this study.
* Having participated in this clinical study.
* History of any chronic degenerative disease, including diabetes and hypertension.
* Presenting active inflammatory or infectious diseases when entering this study.
* Presenting unresolved lesions or trauma when entering this study.
* History of any ocular surgery.
* History of any surgery, non-ocular, within the previous 3 months of entering this studies.
* Being or having an direct family member (spouse, parent/legal guardian, sibling, etc) as employee of the investigation site or the sponsor, who participates directly in this study.

Ages: 18 Years to 35 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 0 (Actual)
Dates: Start 2023-02-01 (Estimated); Primary Completion 2023-03-31 (Estimated); Study Completion 2023-04-24 (Actual)

PRIMARY OUTCOMES:
Incidence of unexpected adverse events | Through Day 21 ± 1 (Safety Call)
  The number of adverse events presented that are not previously described / known for the active substance in this pharmaceutic form and concentration.
Incidence of photophobia | Through Day 21 ± 1 (Safety Call)
  The number of cases of photophobia.

SECONDARY OUTCOMES:
Pupillary Diameter | Days: 1 (Basal Visit), 7 ± 1 (Visit 1), 16 ± 1 (Final Visit)]
  Change of pupillary diameter after exposure to the investigation product.
Incidence of expected adverse events | Through Day 21 ± 1 (Safety Call)
  The number of adverse events presented that are previously described / known for the active substance in this pharmaceutic form and concentration.
Measurement of the change in best near corrected visual acuity (BNCVA) | Time Frame: Days: 1 (Basal Visit), 7 ± 1 (Visit 1), 16 ± 1 (Final Visit)
  The change in BNCVA after exposure to investigation product, compared to basal value.

OTHER OUTCOMES:
Measurement of the change in best corrected visual acuity (BCVA) | Days: 1 (Basal Visit), 7 ± 1 (Visit 1), 16 ± 1 (Final Visit)
  The change in BCVA after exposure to investigation product, compared to basal value.
Changes in intraocular pressure (IOP) | Days: 1 (Basal Visit), 7 ± 1 (Visit 1), 16 ± 1 (Final Visit)
  The change in IOP after exposure to investigation product, compared to basal value.
Incidence of corneal and conjunctival staining | Days: 1 (Basal Visit), 7 ± 1 (Visit 1), 16 ± 1 (Final Visit)]
  Presence of corneal and conjunctival staining with fluorescein and lissamine green after exposure to investigation product.
Measurement of vital signs (blood pressure) | Days: 1 (Basal Visit), 7 ± 1 (Visit 1), 16 ± 1 (Final Visit)
  The change in blood pressure after exposure to investigation product, compared to basal value.
Measurement of vital signs (heart rate) | Days: 1 (Basal Visit), 7 ± 1 (Visit 1), 16 ± 1 (Final Visit)
  The change in heart rate after exposure to investigation product, compared to basal value.
Value of the ocular comfort index (OCI) questionnaire | Days: 1 (Basal Visit), 16 ± 1 (Final Visit)
  The change ocular comfort index (OCI) questionnaire results after exposure to investigation product, compared to basal value.

IPD SHARING:
Plan to Share IPD: No